CLINICAL TRIAL: NCT01664663
Title: Phase II Randomized Study on Locally Advanced Non Small Cell Lung Cancer Escalated Dose on Individual Basis Treatment With Radiochemotherapy
Brief Title: Phase II Randomized Study on Locally Advanced NSCLC Escalated Dose on Individual Basis Treatment With Radiochemotherapy
Acronym: PLANET
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Safety analysis showed increased grade 5 toxicity in experimental arm.
Sponsor: Ass. Prof. Jan Nyman (Network)
Responsible Party: Sponsor-Investigator, Ass. Prof. Jan Nyman, Assosiated professor Jan Nyman, Department of Oncology, Sahlgrenska University Hospital, Gotenburg , Sweden, Swedish Lung Cancer Study Group
Organization: Swedish Lung Cancer Study Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLANET
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Non Small Cell Lung Cancer; Locally Advanced Disease
Keywords: Radiotherapy; Dose escalation; Normal tissue constraints; Locally advanced disease; Good performance status
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A:Standard radiochemotherapy (Active Comparator): Radiotherapy with 2 Gy per fractions 5 fractions a week to 68 Gy to the planning target volume. Three courses of cisplatin 75 mg/m2 day 1and vinorelbine 25 mg/m2 day 1+8. Two courses concomitant with radiation.
  Interventions: Radiation: Standard radiochemotherapy to 68 Gy
- Arm B Escalated radiochemotherapy (Experimental): Radiotherapy with 2 Gy per fraction 5 or 6 times a week to 68-84 Gy to the planning target volume due to normal tissue tolerance constraints. Dose to lung tissue, esophagus and spinal cord will be considered. Three courses of cisplatin 75 mg/m2 day 1 and vinorelbine 25 mg/m2 day 1+8 will be given, two courses concomitant with radiation.
  Interventions: Radiation: Dose escalated radiochemotherapy up to 84 Gy

INTERVENTIONS:
Radiation: Standard radiochemotherapy to 68 Gy
  Arms: Arm A:Standard radiochemotherapy
Radiation: Dose escalated radiochemotherapy up to 84 Gy
  Arms: Arm B Escalated radiochemotherapy

SUMMARY:
The purpose of this study is to examine the valu of individually dose escalated radiotherapy compared with a standard dose of radiotherapy combined with standard concomitant chemotherapy for patients with locally advanced non small cell lung cancer (stage III) with good performance status.

DETAILED DESCRIPTION:
This is an open label, multicentre phase II trial of individually escalated radiotherapy up to 84 Gy due to normal tissue dose constraints combined with standard concurrent chemotherapy (cisplatin-vinorelbine) compared to standard dose radiotherapy (68 Gy) combined with the same chemotherapy. There are restrictions due to lung function, performance status and pre-treatment weight loss. The main endpoint is progression free survival and additional endpoints are local control, overall survival, toxicity quality of life and relapse pattern.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of NSCLC stage IIIA-B.
* Nonresectable or medically inoperable patients.
* No prior chemo- or radiotherapy for NSCLC.
* PS 0-1.
* FEV1 > 1 l or > 40% and CO diffusion capacity > 40%.
* Patient compliance and geographic proximity that allow adequate follow-up.
* Adequate bone marrow reserve: WBCC >3.0, platelets >100, haemoglobin > 100.
* Written informed concent.
* Effective use of contraception.

Exclusion Criteria:

* Excessive weight loss within 6 months (> 10%).
* Supraclavicular nodes.
* Apical tumors-pancoast.
* T4 tumors with separate manifestations in different lobes.
* Evidence of active serious infections.
* Inadequate liver function.
* Inadequate kidney function.
* Pregnancy.
* Breast feeding.
* Serious concomitant systemic disorder.
* Second primary malignancy the last 5 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-09; Primary Completion 2013-11 (Actual); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 36 monts after randomization

SECONDARY OUTCOMES:
Numbers of patients without progression of locoregional disease | 36 months after randomization
  Measured with CT-scan according to the RECIST criteria for response

OTHER OUTCOMES:
Overall survival | 36 months after randomization
Numbers of patients with adverse events | Up to 36 months after randomization
  According to CTC version 4.0
Quality of life | Up to 36 months after randomization
  Measured by questionaires, EORTC QLQ 30 + LC 14

CONTACTS AND LOCATIONS:
Overall Officials: Jan Nyman, Ass. prof, Principal Investigator — Swedish Lung Cancer Study Group
Locations (3):
- Sweden (3):
  - Department of Oncology, Norrlands Universitetssjukhus, Umeå, Norrland
  - Department of Oncology, Karolinska University Hospital, Stockholm, Stockholm County
  - Department of Oncology, Sahlgrenska University Hospital, Gothenburg, Västra Götaland County

REFERENCES:
- [Derived] Hallqvist A, Bergstrom S, Bjorkestrand H, Svard AM, Ekman S, Lundin E, Holmberg E, Johansson M, Friesland S, Nyman J. Dose escalation to 84 Gy with concurrent chemotherapy in stage III NSCLC appears excessively toxic: Results from a prematurely terminated randomized phase II trial. Lung Cancer. 2018 Aug;122:180-186. doi: 10.1016/j.lungcan.2018.06.020. Epub 2018 Jun 18. PMID 30032828